

# HUMAN SUBJECT RESEARCH PROTOCOL-FORM I

**NOTE:** For the purpose of this Form, Mass. Eye and Ear (MEE) include the Massachusetts Eye and Ear Infirmary (MEEI), and Schepens Eye Research Institute, Inc. (SERI). MEEI is a HIPAA-covered entity; SERI is not considered a covered entity.

| DATE: 10/06/14 |
|---|
| <b>TITLE OF PROJECT:</b> Prophylactic antibiotics after functional endoscopic sinus surgery: a randomized, double-blind placebo controlled trial |
| PRINCIPAL INVESTIGATOR: Eric Holbrook |
| FUNDING SOURCE: Dr. Holbrook / Dr. Gray |
| TOTODITO SOURCE. Di. Holotook / Di. Glay |
| 1) Does your research involve the following? Check all that apply: |
| Use of investigational drugs or biologics |
| Use of investigational devices |
| Use of human embryonic stem cells |
| Use of rDNA, microbiological agents, gene transfer, transplantation of animal tissues |
| 2) Is this study a Clinical Trial? XES NO |
| <i>IF YES</i> , submission of an industry-sponsored protocol or SUPP M is required. If no, SUPP N should be |
| submitted. |
| <b>2b)</b> Who will register the study with <u>clinicaltrials.gov</u> ? |
| ☐ This is a Phase I or a pilot study-registration is not required ☐ Sponsor ☐ PI ☐ |
| other:Already registered - NCT01919411 |
| 2) Provide a bai of assessment of the assessment of the leasure of the term have been been assessment of the second of the secon |
| 3) Provide a brief summary of the proposed research (in language that can be understood by a non-scientist): |

RESPONSE: Functional endoscopic sinus surgery (FESS) is a commonly performed procedure in the United States to treat chronic rhinosinusitis. Common practice is to prescribe prophylactic antibiotics postoperatively. This is similar to the long tradition of prophylactic antibiotics after tonsillectomy. The American Academy of Otolaryngology - Head and Neck Surgery recently strongly recommended against prophylactic antibiotics after tonsillectomy. In this light, this study would demonstrate the lack of need for antibiotics after FESS. Currently Dr. Holbrook does not prescribe antibiotics except when evidence of active infection was found during surgery. Dr. Gray currently prescribes antibiotics. This study would prospectively compare the two groups in a randomized fashion. Two previous studies have been performed (Jiang et al. Postoperative antibiotic care after functional endoscopic sinus surgery. Am J Rhinol 22, 608-612, 2008); (Albu, et al. Prophylactic antibiotics in endoscopic sinus surgery: A short follow-up study. Am J Rhinol 24 306-309, 2010.) These studies were both randomized, placebo controlled prospective studies. Albu et al found that amoxicillin/clavulanate improved the outcome in the "early blood crust healing" and the endoscopic score was improved. Jiang et al. showed that amoxicillin/clavulanate did not not improve short term outcomes of FESS. Both studies were limited by a lack

of a prospective instrument to evaluate symptoms. We plan to use the Sinonasal outcomes test -22 (SNOT-22), which is a validated quality of life intrument in sinusitis.

4) What is the estimated completion date? (MM/YYYY)

**RESPONSE: 06/2015** 

Who specifically (name, title, and department) is going to perform the coordinator function? Discuss his/her relevant qualifications (training, education, experience):

The PI, Dr. Holbrook, has assumed coordinator function. He has had experience and training through the Harvard Catalyst education offerings in clinical studies.

- Who is going to supervise the study coordinator(s)? When applicable, indicate if support and oversight will be provided by the Ophthalmology Clinical Research Office (OCRO).
- **6b)** Describe the PI's plan to provide adequate training, and supervision (e.g., regular meetings, training opportunities):

Dr. Holbrook will be supervising all aspects of the study and meets regularly (weekly) with Dr. Gray on matters of enrollment, patient compliance, and monitoring of adverse events.

Delegation of Significant Study-Related Tasks- If non-physicians are tasked to assess clinical response to an investigational therapy, provide medical care to subjects during the course of the study, assess inclusion/exclusion criteria, and evaluate adverse events, list their names in the table below and complete:

| Name | Delegated Tasks | Qualifications- Licensing, or<br>Certification | Training |
|---|---|---|---|
| Dr. Holbrook / Dr. Gray | Enrollment, follow-up,<br>evaluation for adverse<br>reactions, data collection | MD | Residency and fellowship training in otolaryngology and rhinology |
| Pharmacy staff (supervised by Dr. Christine Finn) | Distribution of study drug | Pharm D | Doctorate in pharmacy |

| 8) | Indicate all MEE sites where research activities occur: |
|----|---------------------------------------------------------|
| | ⊠ Boston-MEEI 243 Charles Street |
| | ☐ Boston Longwood Medical Area – 800 Huntington Ave |
| | Boston-SERI 20 Staniford St. |
| | ☐ Braintree - 250 Pond St |
| | Concord - 54 Baker Ave Ext |
| | Duxbury - 20 Tremont St, Route 3A |
| | East Bridgewater - 400 N. Bedford St |

| | Stoneham - One | Washington St<br>ongress St, Crown Col<br>e Montvale Ave<br>ina Consultants-3 Woo | · | | |
|---|---|---|---|---|---|
| 9) | Are there any non- | MEE sites involved in | this stu | dy? 🗌 YES 🔀 NO | (If NO, skip to question 11) |
| <i>IF YE</i> 10) | | site or coordinating cer | | YES NO | occur, and the status of IRB |
| 10) | review at each site | | s for M | EE to serve as the IRB of | record for all study sites (cede |
| | Non-MEE | Sites | IRB | Review Status (i.e., review p | ending, approved, seeking cede<br>ew) |
| | | SURIFO | T INI | FORMATION | |
| | | SOBJEC | | ORMITON | |
| 11) | | please indicate age rar<br>tal number for the stud | | der, total number of subje | ects to be enrolled at MEE, |
| | | Age Range | | Total Number at MEE | Total Number for the Study (if multi-site) |
| Adults<br>Childre | (over 18) | 18- no limit<br>NA | | 0 | 140 |
| (under | | INA | | U | |
| 12) <i>IF YE</i> | Is a gender being e | xcluded from this stud | y? [ | YES NO | |
| Respo | nse: | | | | |
| 13) | 1 1 | ons that may/will be en<br>ay be asked to provide | ` | | the study) below. For some |
| | Pregnant Women | | | | |
| | Employees/Staff of | f MEEI or SERI-please | e specify | y: | |
| | Healthy Controls | | | | |

| | Students/ Residents/ Fellows or other trainees |
|---|---|
| | Children |
| | Prisoner |
| | Non-English Speaking Subjects |
| | Adults with Decisional Impairment- If checked, please describe below the type and range of decisional impairment and a rationale for why it is necessary to include adults with decisional impairment: |
| | Other Populations with Potentially Diminished Capacity (i.e., socially, educationally, economically disadvantaged, elderly, terminally ill) - If checked, specify population below and describe what additional safeguards will be in place to protect the rights and welfare of these subjects: |
| speakii | <b>ONSE:</b> We have enrolled approximately 25 patients so far. We would prefer to enroll non-english ng patients. We are aware of the new IRB protocol regarding non English speaking patients' consent. buld like to apply for the "short-form" consent process in order to continue to enroll non-English speaking es. |
| 14) | Explain how the Investigator has access to a population that would allow recruitment of the required number of subjects within the proposed timeframe: |
| RESP | ONSE: Dr. Holbrook and Dr. Gray both have busy rhinology practices from which to enroll patients. |
| 15) | If subjects are recruited from the investigator's patient population or MEE/SERI employees will be recruited, describe what measures are taken to minimize coercion or undue influence: |
| subject | ONSE: The investigators discuss with the patient the voluntary nature of the study, and the fact that the ts can withdraw at any time from the study. Also it is discussed with the patient that by not enrolling they affect their clinical care at all. |
| | SUBJECT SCREENING/RECRUITMENT |
| 16) | Describe any screening methods used to determine eligible subjects (i.e., search of medical records or recruitment databases, completion of screening tests, response to interview questions, etc.): |
| determ<br>decide | ONSE: Patients will be recruited by Dr. Gray and Dr. Holbrook in their clinics from patients that are nined to be candidates for endoscopic sinus surgery and have agreed to undergo surgery. The patient will to undergo surgery first, and will then be asked to participate in the study. A script to be used for oral ion in the study is provided in the application packet. |
| | Is <u>protected health information</u> accessed during the screening process? YES NO S, specify the information system(s) and the location of the database(s) you will be accessing during the ing process: |
| SCICCIII | ing process. |

| RESPONSE: LMR is accessed for patients' clinical information. This is accessed in the MEEI sinus center. |
|---|
| 18) Is protected health information recorded during the pre-screening process? YES NO IF YES, list the identifiers that are recorded prior to obtaining consent: |
| RESPONSE: |
| Describe the recruitment process (the process by which potential subjects are informed about the availability of the research), who is responsible for recruitment, and how (i.e., use of flyers, advertisements, letters, and oral scripts, etc.) and when subjects will be recruited: |
| RESPONSE: Patients will be recruited by Dr. Gray and Dr. Holbrook in their clinics from patients that are determined to be candidates for endoscopic sinus surgery and have agreed to undergo surgery. The patient will decide to undergo surgery first, and will then be asked to participate in the study. A script to be used for oral invitation in the study is provided in the application packet. |
| 20) Does the recruitment strategy involve contacting individuals multiple times? YES NO IF YES, describe the frequency and in what manner individuals will be contacted: |
| RESPONSE: |
| 21) Are you using email to recruit subjects? |
| RESPONSE: |
| 22) Will fliers, letters and/or brochures be posted, mailed or otherwise distributed? YES NO IF YES, please describe how each document will be used: |
| RESPONSE: |
| <b>NOTE:</b> HIPAA does not permit non-MEE physicians to disclose patient information to Mass. Eye and Ear for research recruitment purposes other than for treatment purposes or pursuant to a HIPAA authorization. Non-MEE physicians may inform their patients of a research study and allow the patients to self-disclose their interest to the study team. |
| Describe whether physician referral is used and whether subjects healthcare providers be notified of their patients' participation in the study? |

RESPONSE: Dr. Gray and Holbrook are rhinology specialists. They are referred patients from community otolaryngologists for management of chronic sinusitis. This involves medical as well as surgical management. Referring otolaryngologists would not be notified of patient participation.

| COMPENSATION/COSTS |
|---|
| Will subjects be paid/offered a recruitment incentive or reimbursed for participating in the research? YES NO |
| <i>IF YES</i> , please describe the amount and type of payment or reimbursement (e.g. parking vouchers) and the proposed method and timing of disbursement and why this is reasonable and non-coercive: |
| Proposer |
| RESPONSE: |
| Will there be any out-of-pocket costs to subjects and/or expenses likely to be covered by their insurance for participating in the study? YES NO |
| IF YES, please specify in detail the costs to subjects and/or their insurance (e.g. co-pays): |
| RESPONSE: The study drug is provided by the pharmacy free of charge. The study medication supplies are charged to the study's cost center by the pharmacy. |
| If applicable, how will the cost of reasonably foreseeable medical care in the event of a research-related injury be covered (e.g., sponsor agreement, likely to be covered by insurance, grant, departmental funds)? |
| RESPONSE: This would be covered by patients' insurance. |
| RISK |
| Risk is the probability and magnitude of harm or discomfort anticipated as a result of participation in the research. Any risks of harm to subjects and/or anticipated discomfort(s) that are reasonably foreseeable, even if unlikely, and the safeguards in place to minimize these risks and discomfort(s) must be identified and discussed below. Risks of harm and discomfort may include: physical harm/discomfort, psychological harm/discomfort, legal harm/discomfort, social harm discomfort, and economic harm. |
| 27) Describe any risks of harm to subjects that are reasonably foreseeable, even if unlikely: |
| These are listed below: 1. amoxicillin/clavulanate arm: From the FDA monograph Gastrointestinal |

Diarrhea, nausea, vomiting, indigestion, gastritis, stomatitis, glossitis, black "hairy" tongue, mucocutaneous candidiasis, enterocolitis, and hemorrhagic/pseudomembranous colitis. Onset of pseudomembranous colitis symptoms may occur during or after antibiotic treatment

# Hypersensitivity Reactions

Skin rashes, pruritus, urticaria, angioedema, serum sickness—like reactions (urticaria or skin rash accompanied by arthritis, arthralgia, myalgia, and frequently fever), erythema multiforme (rarely Stevens-Johnson syndrome), acute generalized exanthematous pustulosis, and an occasional case of exfoliative dermatitis (including toxic epidermal necrolysis) have been reported. These reactions may be controlled with antihistamines and, if necessary, systemic corticosteroids. Whenever such reactions occur, the drug should be discontinued, unless the opinion of the physician dictates otherwise. Serious and occasional fatal hypersensitivity (anaphylactic) reactions can occur with oral penicillin.

### Liver

A moderate rise in AST (SGOT) and/or ALT (SGPT) has been noted in patients treated with ampicillin-class antibiotics but the significance of these findings is unknown. Hepatic dysfunction, including increases in serum transaminases (AST and/or ALT), serum bilirubin, and/or alkaline phosphatase, has been infrequently reported with Augmentin. It has been reported more commonly in the elderly, in males, or in patients on prolonged treatment. The histologic findings on liver biopsy have consisted of predominantly cholestatic, hepatocellular, or mixed cholestatic-hepatocellular changes. The onset of signs/symptoms of hepatic dysfunction may occur during or several weeks after therapy has been discontinued. The hepatic dysfunction, which may be severe, is usually reversible. On rare occasions, deaths have been reported (less than 1 death reported per estimated 4 million prescriptions worldwide). These have generally been cases associated with serious underlying diseases or concomitant medications.

#### Renal

Interstitial nephritis and hematuria have been reported rarely. Crystalluria has also been reported

### Hemic and Lymphatic Systems

Anemia, including hemolytic anemia, thrombocytopenia, thrombocytopenic purpura, eosinophilia, leukopenia, and agranulocytosis have been reported during therapy with penicillins. These reactions are usually reversible on discontinuation of therapy and are believed to be hypersensitivity phenomena. A slight thrombocytosis was noted in less than 1% of the patients treated with Augmentin. There have been reports of increased prothrombin time in patients receiving Augmentin and anticoagulant therapy concomitantly.

# Central Nervous System

Agitation, anxiety, behavioral changes, confusion, convulsions, dizziness, insomnia, and reversible hyperactivity have been reported rarely.

#### Miscellaneous

Tooth discoloration (brown, yellow, or gray staining) has been rarely reported. Most reports occurred in pediatric patients. Discoloration was reduced or eliminated with brushing or dental cleaning in most cases.

## 2. Placebo Arm:

The main theoretical risk from not giving antibiotics post operatively would be a risk of postoperative infection. This would manifest as sinusitis-like symptoms. Worst case scenario would result in complications of sinusitis (orbital infection, meningitis, brain abscess). These complications are rare, and Dr. Holbrook has not experienced them while not giving routine postoperative antibiotics as is his usual practice.

# 3. Privacy:

| remove personal identifying information from the research data. Data will be secured under a password protected computer in a locked office of the PI. |
|---|
| 28) If applicable, describe any group harms (i.e., research that focuses on a specific group or population): |
| RESPONSE: NA |
| Do you anticipate any circumstances in which a "breach of confidence" associated with a mandated disclosure (e.g. reporting abuse to authorities) may occur as part of this study? |
| RESPONSE: No we do not anticipate a breach of confidence |
| 30) In the view of the PI, what risk classification (taking into consideration the probability and magnitude of harm) is appropriate for the proposed research? ☐ Minimal Risk ☐ Greater than Minimal Risk ☐ Unknown Minimal risk means the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests. |
| Please explain why you feel this category is appropriate based on the definition above (when more than minimal risk describe the likelihood and seriousness of such risks): |
| RESPONSE: In patients that are randomized to receive post operative antibiotics, there is a risk of adverse reaction to augmentin as detailed above. For patients that are randomized to placebo, there is a risk of post operative infection as detailed above as well. We believe the study is low risk to participants, however as defined above, it is more than the risk encountered in daily life. |
| 32) What provisions are in place to minimize harm or discomfort? |
| RESPONSE: Patients are seen one week after surgery to undergo endoscopic evaluation to ensure that the patient is healing well without evidence of infection. At all times during the day they can call the sinus center to speak to a nurse if they have any concerns. At night there is a resident on call to answer questions and the MEEI ED is always open. |
| ALTERNATIVES |

Describe any alternatives, especially other treatment(s) that are available to potential patients outside of the research:

8

33)

RESPONSE: If patients do not elect to enroll in the study, they would receive standard post-operative care. They would be prescribed antibiotics at the discretion of the surgeon.

| BENEFITS | R | $\mathbf{E}$ | V | $\mathbf{E}$ | $\mathbf{F}$ | $\Gamma$ | S |
|----------|---|--------------|---|--------------|--------------|----------|---|
|----------|---|--------------|---|--------------|--------------|----------|---|

| 34) | Are there any potential direct benefits to individual subjects related to the research? YES NO |
|---|---|
| | <b>S</b> , please explain (address whether these benefits (e.g., clinical, therapeutic) would be available to its outside of the research): |

# **RESPONSE:**

Explain the potential benefits to science, and/or society (indirect benefits) which may accrue as a result of this research:

RESPONSE: Antibiotic resistance is growing in the world, and this study may provide prospective, randomized data that antibiotics do not result in a benefit to patients. Hopefully surgeons would stop giving postoperative antibiotics, and decrease the risk of side-effects from antibiotics (allergic reactions, clostridium dificile infection, GI upset, etc) to future patients. Also health care costs would be decreased by reducing antibiotic prescriptions.

**36)** If more than minimal risk, address how risks relate to benefits:

RESPONSE: While not "minimal risk", the risk to patients is low, as detailed above. Many patients have adverse reactions to antibiotics, and if this study shows that the outcomes of patients undergoing sinus surgery without antibiotics are not worse, then hopefully less patients will be prescribed antibiotics.

# CONSENT PROCESS

Describe the consent process in detail. Include who specifically will be obtaining consent, describe their knowledge/experience in obtaining consent from research subjects, and include the location where study information will be exchanged, how (consent form, orally, information sheet, etc.) information is being conveyed to subjects, and when the consent will be obtained (e.g. during pre-surgical visit, about one week before the screening visit):

RESPONSE: Consent will be obtained by Dr. Gray, Dr. Meier or Dr. Holbrook in the clinic during the subject's preoperative visit in the MEEI sinus center. There is a formal consent form that is signed by patients and an oral script (these are on IRBNET). Subjects can think about the study and opt out of randomization at the time of surgery (usually 2-4 weeks elapse between preoperative visit and surgery).

| 38) | Indica | te which of the following consent procedures you are contemplating for this research: |
|---|---|---|
| | $\boxtimes$ | Written consent form |

| | Short form process (only appropriate for minimal risk studies) * If checked, answer question 42 below. |
|---|---|
| | Assent from adults with diminished decision-making capacity *If checked, provide justification below: |
| | Assent from children and parental permission |
| | Oral consent or implied consent (e.g. completing a survey) *If checked, provide justification based on 45 CFR 46.117(c) below: |
| | Requesting a waiver of informed consent from the HSC *If checked, provide justification based on 45 CFR 46.116(c) and (d) below: |
| RESPONSE | :<br>: |

39) Describe any foreseeable circumstances and/or reasons under which the subject's participation in the research may be terminated:

RESPONSE: If the patient does not want to participate further then they may opt out at any time during the study.

40) How is subject comprehension assessed initially and throughout the consent process? Is the manner in which information is presented appropriate for the population? In cases where subject comprehension is severely limited what special provisions have been made (is there a third party involved in the consent process)? Discuss below:

RESPONSE: The investigators will describe the study according to the oral script and ask the patient if they understand everything that has been explained to them. We will ask them if they have any questions and answer them to their satisfaction. If the patients' comprehension is severely limited then we will not include them in the study.

41) If the research-related intervention or interaction will occur on the same day that the subject initially receives information about the study, justify why this is appropriate/necessary:

RESPONSE: It will not be on the same day, patients will be enrolled at their post operative visit.

Describe additional provisions in place for non-English speaking subjects (view <u>guidance</u>), including the availability/presence of translators (fluent in both English and the subject's spoken language) during the consent process and the translation of consent documents in a language understandable to them (when consent documents are translated all translated versions must be accompanied by an attestation from the translator) **OR** justify why non-English speaking subject are being excluded from the research:

RESPONSE: We would like to apply for use of the short form consent process for patients that do not speak English. We have used translators for patients that are not English speakers previously.

43) How will literacy be assessed? If subjects cannot read the consent form, describe the process for providing information to these subjects (i.e., reading the information aloud) and for documenting consent, including whether or not the short form (45 CFR 46.117(b) (2)) process will be utilized:

RESPONSE: This has not come up in the year of our trial. We would ask subjects if they understand the written consent form. If they are not literate, then we would use the oral script and document their understanding.

For Ophthalmology related studies, describe if the cohort is capable of reading the consent form and if not, describe exacerbating factors (visual impairment, eyes dilated at the onset of the study, etc.). In these cases, describe additional measures you will take to ensure comprehension of study-related information to promote informed decision-making by the subject:

**RESPONSE: NA** 

45) For Otology related studies, describe if the cohort is capable of comfortably hearing the Investigator during the consent process and if not, describe exacerbating factors (hearing aid, cochlear implant, hearing impaired, etc.). In these cases, describe additional measures you will take to ensure comprehension of study-related information to promote informed decision- making by the subject:

**RESPONSE: NA** 

## INCIDENTAL FINDINGS

Is there a possibility of clinically significant incidental findings (information relating to previously undiagnosed medical or psychiatric conditions) being discovered during research procedures?

YES

NO

*IF YES*, please outline the plan for addressing incidental findings (i.e., contacting the subject's primary care provider, referral etc.) including if and how subjects will be informed:

**RESPONSE:** 

# DISSEMINATION OF RESULTS

Describe any plans to share research results with subjects, this may include sharing individual results and/or aggregate results and may also serve as an opportunity to follow-up with subjects and **thank** them for participating in the research, particularly in cases where there is no direct benefit to the subject. If there are no plans to share results explain why this is not feasible, appropriate or applicable to this research:

RESPONSE: We would plan on disseminating the final publication paper to the subjects with a note of thanks when the research is completed.

| 48) | How will results be published, and in what form (i.e., subjects will not be individually identifiable in publications): |
|---|---|
| RESPONSE: Results will be published in an otolaryngology peer-reviewed journal. There will be no identifiable information in the publication. | |
| PRIVACY/CONFIDENTIALITY | |
| Insofar as they apply, investigators are required to adhere to <u>MEE Information Security Policies and Procedures</u> . Therefore, research protocols must be designed in accordance with these requirements. On occasion the HSC may require additional provisions related to the use and security of research data. The HSC | |

evaluates the collection and use of data based on the minimum necessary standard, the data necessary to satisfy the purposes of the research to carry out research-related activities. The HSC may require that when a research project collects personally identifiable, sensitive information that the PI obtain a Certificate of Confidentiality.

49) Describe the provisions in place to respect the privacy of subjects throughout the research:

RESPONSE: For each subject in the study, a unique identification number will be generated, this number will be used with their study responses and all results from the study. A list linking patients' names, MRN and unique ID will be created and stored on a password-protected computer only accessible by the PI. The survey responses with the unique identifiers will be locked in the PI's office. Only the PI will have access to this list. Pharmacy will have access only to the unique ID, and will be in charge of randomization.

| 50) Check all identifiers that will be obtained by investigate | ors for the purposes of this study. |
|---|---|
| <ul> <li>Name</li> <li>Social Security Number</li> <li>Medical Record Number</li> <li>Address by Street Location</li> <li>Address by Town/City/Zip Code</li> <li>Health Plan Beneficiary Number</li> <li>Certificate/License Number</li> <li>Full Face Photographic Image</li> <li>Elements of Dates except Year (Admission/Discharge Date</li> <li>Vehicle ID Number and Serial Number Including License F</li> <li>Medical Device Identifiers and Serial Number</li> <li>Biometric Identifiers (e.g. finger or voice prints, retinal ima</li> <li>None of the listed identifiers will be recorded as part of this</li> </ul> | Telephone Number Fax Number Email Address Web URLs Internet Protocol (IP) Address Account Number Ages over 89 The system of Birth or Death Plate Number The system of Birth or Death The system of Birth or Death The system of Birth or Death |
| Other unique identifiers or code that can be used to identify the participant: | |

51) Investigators should only obtain the minimum data necessary to achieve research goals. Please justify why the data you are obtaining is the minimum necessary:

RESPONSE: We need the patients' names, date of birth, and MRN to identify patients. A unique number will be generated that will deidentify the patients to the pharmacy.

| 52) | Will data about individual subjects be collected from sources outside of Mass. Eye and Ear? YES NO |
|---|---|
| <i>IF YES</i> , list each source (include if the source is considered a covered entity), the data collected, and any agreements in place to allow transfer of this data: | |
| RESP | ONSE: |
| 53) | Sensitive information includes (but is not limited to) information relating to sexual attitudes, preferences, or practices; information relating to the use of alcohol, drugs, or other addictive products; information pertaining to illegal conduct; information that, if released, might be damaging to an individual's financial standing, employability, or reputation within the community or might lead to social stigmatization or discrimination; information pertaining to an individual's psychological well-being or mental health; and genetic information or tissue samples. |
| | Will this research collect sensitive information? |
| IF YE | S, list the data that will be collected and provide a rationale under the <i>minimum necessary</i> standard: |
| DECD | PONSE: |
| KESI | UNSE: |
| Has a Certificate of Confidentiality been sought for this research? YES NO | |
| <i>IF YES</i> , include a copy of the certificate at the time of submission or provide information related to the status of your application | |
| <i>IF NO</i> , justify your response below: | |
| 55) | Please indicate the specific safeguards in place to protect the confidentiality of subject data: |
| Administrative Safeguards: | |
| ⊠ YE | ES NO Each member of the study team has completed Mass. Eye and Ear Privacy Training and Information Security Awareness Training and this training is up to date. |
| ⊠ YE | Paper files, electronic data, computing devices and storage media will be safeguarded in accordance with Mass. Eye and Ear Privacy and Information Security policies and procedures, including, but not limited to the safeguards more specifically identified below: |
| Physical Safeguards: | |
| ⊠ YE | ES NO N/A Paper files will be locked in cabinets when not in use |
| ☐ YE | ES NO N/A Paper files will be protected from inappropriate access when in use |

| ☐ YES ☐ NO ☑ N/A | Mobile computing devices and storage media will be locked in cabinets when not in use |
|---|---|
| ≥ YES □ NO □ N/A | Computing devices will be protected from inappropriate access when in use |
| Yes No N/A | Research data will be coded using a subject identification number that does not include the subject's initials and is not derived from the subject's identifiable information. |
| | <b>IF YES:</b> The key linking the subject identification number to the subject's identifiable information is available only to the following study team members: |
| | <ul> <li>✓ Mass. Eye and Ear PI</li> <li>✓ Other Mass. Eye and Ear study team members</li> <li>✓ External investigator</li> <li>✓ External sponsor</li> </ul> |
| ⊠ Yes □ No | The key will be stored separately and in a locked cabinet (if paper) |
| ⊠ Yes □ No | The key will be stored separately and on a password protected network drive with access limited to those people identified above |
| | Technical Safeguards: |
| ⊠ YES □ NO | Electronic data will be stored on Mass. Eye and Ear network folders for which access is limited to authorized members of the study team only |
| ⊠ YES □ NO | To the extent that electronic data is collected on the hard drive of a computing device, it will be promptly and securely transferred to a secure folder within the Mass. Eye and Ear network |
| ⊠ YES □ NO | Mobile devices (including but not limited to laptops, tablet computers, smart phones, external hard drives and USB drives) containing electronic data will be encrypted |
| ☐ YES ⊠ NO | Remote access to electronic data will be gained through Information Systems |
| ☐ YES ⊠ NO | Electronic data will be encrypted when transmitted outside of Mass. Eye and Ear |
| Please describe any additional safeguards that will be used to protect the study data and explain any "No" responses: | |
| RESPONSE: We will not use remote access, and we will not send data outside of MEEI. | |
| Will data that identifies individual subjects be disclosed to parties outside of Mass. Eye and Ear (e.g. sponsor and/or coordinating center, research registry) for purposes of the research? YES NO | |

| IF YI | ES, list the parties and explain how and what information will be shared: |
|---|---|
| RESPONSE: | |
| 55) | WI 'II 114 ' 11' 4 ' 1' C 1 4 C 1 4 A ACET |
| 57) | Where will research data, including the signed informed consent form and assent be stored (e.g., MEEI medical record, research record, etc.). |
| | * |
| RESI | PONSE: In the MEEI Sinus center under lock and key. |
| 58) | Please provide the plan for destroying identifiers (at the earliest opportunity as consistent with the research plan) or provide a health or research justification for retaining identifiers. For protocols subject to future and secondary data analysis, provide justification for not destroying identifiers permanently and explain plans for future use (i.e., establishment of a data or specimen repository): |
| | PONSE: When the research is complete, we will destroy all identifiable information by following I protocols. |
| WIE | i protocois. |
| | CONFLICTS OF INTEREST |
| t. | |
| If the research involves any of the following: 1) for-profit sponsor or funding source; 2) a marketed drug, device, or other technology; or a drug, device, or other technology in development; or 3) a new technology, software, or therapeutic approach, all investigators are required to complete and submit (at the time of initial submission and thereafter in accordance with the policy) a Conflict of Interest in Research: Project-Specific Disclosure (SUPP L) in accordance with the HSC Conflicts of Interest: Clinical Research policy. Please refer to the policy and SUPP L for further guidance on disclosure and submission requirements. FAQ guidance on this topic is also available. | |
| 59) | Does the research involve (check all that apply): |
| | For-profit sponsor or funding source? \(\begin{aligned} \text{YES} & \simeq \text{NO} \end{aligned}\) |
| | Marketed drug, device, or other technology; or a drug or device, or other technology in development?<br>XES NO |
| We are using amoxicillin / clavulinate as the study drug. This drug is generically available in the US. We are not seeking a new indication for this already FDA approved medication. | |
| | New technology, software, or therapeutic approach? |